CLINICAL TRIAL: NCT04064489
Title: Thromboembolic Risk Stratification by TRIP Score (Cast) to Guide Physicians in Preventive Treatment Prescriptions for Patients With Lower Limb Trauma Requiring Brace or Casting.
Brief Title: Thromboembolic Risk Stratification by TRiP(Cast) Score to Guide Physicians in Preventive Treatment Prescriptions for Patients With Lower Limb Trauma Requiring Brace or castING.
Acronym: CASTING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Centre Hospitalier de Cholet (Other); Centre Hospitalier de Saint-Brieuc (Other); Bichat Hospital (Other); Hôpital Cochin (Other); University Hospital, Toulouse (Other); University Hospital, Grenoble (Other); Centre Hospitalier Régional d'Orléans (Other); Poitiers University Hospital (Other); Nantes University Hospital (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); University Hospital, Tours (Other); CHU Rennes - Hopital Pontchaillou (Other); Centre Hospitalier le Mans (Other); Centre Hospitalier d'Agen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 49RC19_0027
Record Dates: First submitted 2019-08-19; First posted 2019-08-22 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Lower Limb Trauma; Venous Thromboembolism; Stratification
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neutral (No Intervention): No specific instructions for prescribing prophylaxis or not
- TRIPscore (Active Comparator): calculation of the TRIPcast score and prescription of prophylactic or not according to the result (score > or = 7 : treatment (low molecular weight heparin or fondaparinux); score < 7 : no treatment)
  Interventions: Other: TRIPscore

INTERVENTIONS:
Other: TRIPscore — TRIPcast score calculation
  Arms: TRIPscore

SUMMARY:
Non-surgical traumas to the lower limbs that require orthopedic immobilisation (plaster or splint) are a frequent reason for going to accident and emergency. Due to venous stasis caused by immobilisation, hypercoagulable states and vascular injuries brought on by the trauma, these patients are at risk of developing VTE. For this reason, it is current practice in France and Belgium for the majority of patients to receive a preventative anticoagulant treatment. However, the benefit of this treatment, which has a considerable cost, is controversial. Contrary to French recommendations, American recommendations from 2012 actually advise against systematic preventative medicine, with prevention appearing to be effective primarily in studies with restrictive inclusion criteria. The most significant randomised controlled study on the subject did not show the benefit of low-molecular-weight heparin (LMWH) on the rate of symptomatic VTE among 1,435 non-selected patients. Therefore, in 2017, the Cochrane meta-analysis concluded that stratification of the risk of thromboembolism is required.

For this purpose, in collaboration with the Dutch team of Nemeth et al. we have recently developed a risk stratification model that takes into consideration the patient's characteristics, the type of immobilisation and the severity of the trauma: the TRiP(cast) score. This score is applied retrospectively to a large cohort and demonstrates excellent prognostic performances (AUC (area under the curve) of 0.74). In addition, when using a <7 limits, it makes it possible to identify a large group of patients at very low risk of developing VTE (negative predictive value: 99.2%).

The aim of the CASTING study is to prospectively demonstrate the reliability and utility of the TRiP(cast) score by showing that patients with orthopaedic immobilisation of a lower limb who are not receiving preventative treatment on the basis of a TRiP(cast) score of <7 have a very low rate of symptomatic VTE, which allows for a significant reduction in prescriptions of anticoagulants in comparison with prior practices.

ELIGIBILITY:
Inclusion Criteria:

* Consultation in one of the emergency department participating in the study,
* Isolated trauma from lower limb,
* Rigid (plaster or resin) or semi-rigid immobilization for an assumed duration of at least 7 days,
* Adults (18 years),
* Affiliated patient or beneficiary of a social security,
* Patient with prior informed consent.

Exclusion Criteria:

* Patient with anticoagulant treatment at the time of trauma,
* Trauma requiring hospitalization of more than 48 hours,
* Co-morbidity(s) requiring hospitalization of more than 48 hours at the time of inclusion,
* Any factor making 90-day follow-up impossible,
* Pregnant, nursing or childbearing patient,
* Patient deprived of liberty by judicial or administrative decision,
* Patient undergoing psychiatric care under duress,
* Patient subject to a legal protection measure,
* Patient unable to give free and informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2123 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Rate of symptomatic venous thromboembolic events (deep vein thrombosis and / or pulmonary embolism) among patients with a TRiP(cast) score < 7 | Day 90
  To demonstrate the reliability and safety of the decision not to implement thromboprophylaxis in patients with orthopedic immobilization for lower extremity trauma and Trip(cast) < 7

SECONDARY OUTCOMES:
Rate of prescription for thromboprophylaxis | Day 1
  comparison between the two period
Rate of symptomatic venous thromboembolic events (deep vein thrombosis and / or pulmonary embolism) (whole population) | Day 90
  comparison between the two period
The rate of complications of preventive anticoagulant treatment (bleeding) | Day 90
  comparison between the two period
The direct cost of preventive anticoagulant treatment when the TRiP(cast) score is applied compared to current practices | Day 90
  treatment, nurse, blood test...cost of care
Physicians' satisfaction using likert's scale | Day 1
  5 level ladder : from totally unsatisfied to totally satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Marie Roy, MD PhD, Study Chair — University Hospital, Angers
Locations (15):
- Clinique Universitaire Saint-Luc, Brussels, Belgium
- France (14):
  - Centre Hospitalier d'Agen, Agen
  - CHU Angers, Angers
  - Centre Hospitalier de Cholet, Cholet
  - Centre Hospitalier Universitaire de Grenoble, Grenoble
  - Centre Hospitalier Le Mans, Le Mans
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Centre Hospitalier d'Orléans, Orléans
  - APHP Bichat, Paris
  - APHP Cochin, Paris
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Centre Hospitalier Universitaire de Rennes, Rennes
  - Centre Hospitalier de Saint-Brieuc, Saint-Brieuc
  - Centre Hospitalier Universitaire de Toulouse, Toulouse
  - Centre Hospitalier Universitaire de Tours, Tours

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available. The study protocol, the Statistical Analysis Plan, Informed consent form will be available immediately following publication. No end date.

REFERENCES:
- [Derived] Douillet D, Penaloza A, Viglino D, Banihachemi JJ, Abboodi A, Helderle M, Montassier E, Balen F, Brice C, Laribi S, Duchenoy T, Vives P, Soulat L, Marjanovic N, Moumneh T, Savary D, Riou J, Roy PM. Targeted prophylactic anticoagulation based on the TRiP(cast) score in patients with lower limb immobilisation: a multicentre, stepped wedge, randomised implementation trial. Lancet. 2024 Mar 16;403(10431):1051-1060. doi: 10.1016/S0140-6736(23)02369-3. Epub 2024 Feb 15. PMID 38368901
- [Derived] Douillet D, Riou J, Thoma M, Moumneh T, Darsonval A, Trinh-Duc A, Hugli O, Chauvin A, Penaloza A, Roy PM. Thromboembolic risk stratification by TRiP(cast) score to rationalise thromboprophylaxis in patients with lower leg trauma requiring immobilisation: a study protocol of the casting stepped-wedge cluster randomised trial. BMJ Open. 2021 Jun 28;11(6):e045905. doi: 10.1136/bmjopen-2020-045905. PMID 34183341